CLINICAL TRIAL: NCT06378489
Title: The Etonogestrel Contraceptive Implant for Treatment of Endometrial Hyperplasia Without Atypia: A Single-arm, Open-label, Longitudinal Study in a Government Hospital in the Philippines
Brief Title: The Use of Etonogestrel Contraceptive Implant as Treatment for Endometrial Hyperplasia Without Atypia: A Cohort Study
Status: Not yet recruiting | Type: Observational
Sponsor: University of the Philippines (Other)
Collaborators: Organon (Industry)
Responsible Party: Sponsor
Other Study IDs: 2022-0346-01
Record Dates: First submitted 2024-04-17; First posted 2024-04-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Endometrial Hyperplasia Without Atypia
Keywords: endometrial hyperplasia without atypia; etonogestrel implant
MeSH Terms: interventions — etonogestrel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Etonogestrel implant — The etonogestrel implant will be inserted on the inner side of the non-dominant upper arm of the patient. Three months after insertion, a repeat transvaginal ultrasound will be performed to document endmetrial thickness and an endometrial biopsy will also be done using the Pipelle to document the histology of the endometrium. If the biopsy showed regression of the hyperplasia, the implant will be left in place for a minimum of 12 months until 3 years. If the repeat biopsy showed non-resolution of the hyperplasia, the patient will be referred to a gynecologic oncologist for further management
  Other Names: Implanon NXT

SUMMARY:
Endometrial hyperplasia without atypia is a condition in which the endometrium (the lining of the uterus) becomes abnormally thick. Although endometrial hyperplasia without atypia is not cancer, it can lead to endometrial cancer in 1-3% of women. This disease is treated by giving progestins. The optimal route, dosage and duration of progestin treatment for endometrial hyperplasia has not yet been determined until now. However, several publications have suggested the use of levonorgestrel releasing IUD as first-line treatment for endometrial hyperplasia without atypia. The other common medications used are the oral progestins medroxyprogesterone (MPA) and norethisterone acetate (NETA).

The etonogestrel implant (Implant NXT) has been approved for contraceptive use by the US FDA in 2006. The mchanism of action of the implant for contraception suggests a potential application for its use in the treatment on hyperplasia. Off-label use of the implant for adrnomyosis, endometriosis and chronic pelvic pain has already been described in various studies. However, its therapeutic effect on endometrial hyperplasia without atypia has not been studied yet. The researchers propose to use the etonogestrel implant (Implant NXT) as novel treatment for endometrial hyperplasia without atypia. The study aims to determine the rate of regression to normal endometrium among patients with endometrial hyperplasia without atypia at 3 and 6 months after insertion of the implant.

ELIGIBILITY:
Inclusion Criteria:

* women aged 18 years old to perimenopause who present with or without abnormal uterine bleeding and who have an endometrial biopsy result which shows endometrial hyperplasia without atypia
* women willing to have the etonogestrel implant (Implant NXT) for the duration of treatment (6-12 months)
* women who wish to retain their uterus

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women aged 18 years old to perimenopause who present with or without abnormal uterine bleeding and who have an endometrial biopsy result which shows endometrial hyperplasia without atypia
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Rate of (resolution) regression to normal endometrium | 3 months after the insertion of the implant
Endometrial thickness (by ultrasound) | At three and six months after insertion of the implant
  Performed by expert sonologist

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Jose D Padilla, MD, Principal Investigator — Philippine General Hospital

IPD SHARING:
Plan to Share IPD: Undecided